## **Table of Contents**

| STATISTICAL ANALYSIS PLAN | 1 |
|---|---|
| 1. INTRODUCTION | 9 |
| 2. OBJECTIVES | 9 |
| 3. OVERALL STUDY DESIGN | 9 |
| 4. IDENTITY O F INVESTIGATIONAL PRODUCT | 14 |
| 5. RANDOMIZATION AND BLINDING | 14 |
| 6. SAMPLE SIZE | 15 |
| 7. STUDY POPULATIONS | 16 |
| Per-Protocol (PP) Population | 16 |
| Pharmacodynamic (PD) Population | 16 |
| Safety Populations | 16 |
| 8. STATISTICAL ANALYSIS METHODS | 17 |
| 8.1 Baseline Characteristics. | |
| 8.1.1 Patient Disposition. | |
| 8.1.2 Demographic and Other Baseline Characteristics | |
| 8.1.3 Medical History | |
| 8.1.4 Concomitant Medications. | 18 |
| 8.2 Pharmacodynamic Equivalence Analyses | |
| 8.2.1 Primary Pharmacodynamic Endpoint | |
| 8.2.2 Population | 19 |
| 8.2.3 PC20 Log Transformation | 19 |
| 8.2.4 NONMEM® Dataset Preparation | 19 |
| 8.2.5 Dose-Scale Approach | 19 |
| 8.2.6 Dose Response Emax Model | 20 |
| 8.2.7 Alternative Approach to the Dose Response Emax Model | 20 |
| 8.2.8 Bootstrap | 25 |
| 8.2.9 Calculation of Confidence Intervals for Frel | 25 |
| 8.2.10 Calculation of Confidence Intervals for Frel | 26 |
| 8.3 Safety Analysis | 26 |
| 8.3.1 Adverse Events. | 26 |
| 8.3.2 Vital Signs | 27 |
| 8.3.3 Physical Exam | 27 |
| 8.3.4 12-lead ECG | 27 |
| 8.3.5 Pregnancy Test. | 28 |
| 8.3.6 Concentration of Methacholine Required to Reduce FEV1 by 20% ( | (PC20) |
| | 28 |
| 8.3.7 Forced Expiratory Volume (flow rate) in 1 second (FEV1) | 28 |

| | 8.3.8 Protocol Deviations | 28 |
|---|---|---|
| | 8.4 Multiple Comparisons | 28 |
| | 8.5 Methods for Handling Missing Data | 28 |
| | 8.6 Interim Analyses. | 28 |
| 9. | TABLE, LISTING AND FIGURE SHELLS | 28 |
| | T16.1.9.1 Summary of Patient Disposition | 30 |
| | T16.1.9.2 Summary of Protocol Deviations | 31 |
| | T16.1.9.3 Summary of Patient's Treatments Included in the Pharmacodynamic Analysis | |
| | | 32 |
| | T16.1.9.4 Summary of Demographic Data and Baseline Characteristics | 33 |
| | T16.1.9.5 Summary of Demographic Data and Baseline Characteristics | 35 |
| | T16.1.9.6 Summary of Demographic Data and Baseline Characteristics | 35 |
| | T16.1.9.7 Summary of Concentration (mg/mL) of Methacholine Required to Reduce | |
| | FEV1 by 20% (PC20) | 36 |
| | T16.1.9.8 Summary of Concentration (mg/mL) of Methacholine Required to Reduce | |
| | FEV1 by 20% (PC20) | 36 |
| | T16.1.9.9 Summary of Concentration (mg/mL) of Methacholine Required to Reduce | |
| | FEV1 by 20% (PC20) | 36 |
| | T16.1.9.10 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 | |
| | second (FEV1). | 37 |
| | T16.1.9.11 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 | |
| | second (FEV1). | 38 |
| | T16.1.9.12 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 | |
| | second (FEV1). | 38 |
| | T16.1.9.13 Overall Summary of Adverse Events | 39 |
| | T16.1.9.14.1 Summary of Frequency of All Adverse Events by System Organ Class | |
| | | 40 |
| | T16.1.9.14.2 Summary of Frequency of Serious Adverse Events by System Organ Class | |
| | | 41 |
| | T16.1.9.15.1 Summary of Frequency of All Adverse Events by Relationship to Study | |
| | Drug | 42 |
| | T16.1.9.15.2 Summary of Frequency of Serious Adverse Events by Relationship to | |
| | Study Drug. | 43 |
| | T16.1.9.16.1 Summary of Frequency of All Adverse Events by Severity | 44 |
| | T16.1.9.16.2 Summary of Frequency of Serious Adverse Events by Severity | 45 |
| | T16.1.9.17 Summary of Vital Signs | 46 |
| | L16.2.1 Listing of Discontinued Subjects | 47 |
| | L16.2.2 Listing of Protocol Deviations | |

| L16.2.3.1 Listing of Subjects Excluded from the Per-Protocol Population | 49 |
|---|---|
| L16.2.3.2 Listing of Subjects Excluded from the Pharmacodynamic Population | 50 |
| L16.2.4.1 Listing of Demographic Data | 51 |
| L16.2.4.2 Listing of Medical History | 52 |
| L16.2.4.3 Listing of Concomitant Medication | 53 |
| L16.2.5 Listing of Dosing | 54 |
| L16.2.6.1 Listing of Methacholine Challenge and Pulse Oximetry | 55 |
| L16.2.6.2 Listing of Methacholine Challenge Stages | 56 |
| L16.2.6.3 Listing of Spirometry Test. | 58 |
| L16.2.7.1 Listing of Adverse Events (Safety Population Randomization Period) | 59 |
| L16.2.7.2 Listing of Adverse Events (Safety Population Screening Period) | 60 |
| L16.2.7.3 Listing of Positive Pregnancy Test Results | 61 |
| L16.2.7.4 Listing of Abnormal Physical Examinations | 62 |
| L16.2.8.1 Listing of Vital Signs | 63 |
| L16.2.8.2 Listing of 12-Lead ECG. | 64 |
| NTF- Tables and Listings Numberings Change | 66 |

#### Albuterol Sulfate Inhalation Aerosol

Protocol / Study No. CLR 17 08/

#### STATISTICAL ANALYSIS PLAN

A Randomized, Single-Dose, Double-Blind, Double-Dummy, Four-Period, Four-Sequence, Four-Treatment, Placebo and Active Controlled, Comparative, Multiple-Center, Crossover-Design, Bronchoprovocation Study to Evaluate the Pharmacodynamic Equivalence of Albuterol Sulfate Inhalation Aerosol, eq 90 mcg base (Sun Pharmaceuticals Industries Limited) to PROAIR® HFA (albuterol sulfate) Inhalation Aerosol, eq 90 mcg base (Teva Respiratory, LLC) in Subjects With Stable, Mild Asthma

Protocol Number: CLR 17 08

#### **Sponsor:**

Sun Pharmaceuticals Industries Limited Formulation Development Department Tandalja, Baroda Gujarat, 390020, India



December 21, 2018

Final Version 1.0

Protocol / Study No. CLR 17 08/

#### SAP FINAL VERSION APPROVALS

A Randomized, Single-Dose, Double-Blind, Double-Dummy, Four-Period, Four-Sequence, Four-Treatment, Placebo and Active Controlled, Comparative, Multiple-Center, Crossover-Design, Bronchoprovocation Study to Evaluate the Pharmacodynamic Equivalence of Albuterol Sulfate Inhalation Aerosol, eq 90 mcg base (Sun Pharmaceuticals Industries Limited) to PROAIR HFA (albuterol sulfate) Inhalation Aerosol, eq 90 mcg base (Teva Respiratory, LLC) in Subjects With Stable, Mild Asthma



■ Sun Pharmaceuticals Industries Limited ■


#### SAP FINAL VERSION APPROVALS

A Randomized, Single-Dose, Double-Blind, Double-Dummy, Four-Period, Four-Sequence, Four-Treatment, Placebo and Active Controlled, Comparative, Multiple-Center, Crossover-Design, Bronchoprovocation Study to Evaluate the Pharmacodynamic Equivalence of Albuterol Sulfate Inhalation Aerosol, eq 90 mcg base (Sun Pharmaceuticals Industries Limited) to PROAIR® HFA (albuterol sulfate) Inhalation Aerosol, eq 90 mcg base (Teva Respiratory, LLC) in Subjects With Stable, Mild Asthma



12/21/2018

■ Sun Pharmaceuticals Industries Limited ■


# Albuterol Sulfate Inhalation Aerosol

Protocol / Study No. CLR 17 08/

# **Revision History**

| VERSION | DATE | DESCRIPTION OF REVISIONS | REVISED<br>BY |
|---|---|---|---|
| Draft 1.0 | September 24, 2018 | New Document | |
| Final 1.0 December 21, 2018 | | Incorporate client's comments and finalize SAP | |

# Albuterol Sulfate Inhalation Aerosol

Protocol / Study No. CLR 17 08/

## **List of Abbreviations and Terms**

| <b>Abbreviation</b> | <u>Term</u> |
|---|---|
| AE | Adverse Event |
| ADaM | Analysis Data Model |
| ANDA | Abbreviated New Drug Application |
| ATS | American Thoracic Society |
| C | Celsius |
| CDISC | Clinical Data Standards Interchange Consortium |
| CRO | Clinical Research Organization |
| ECG | Electrocardiogram |
| eCRF | electronic Case Report Form |
| eCTD | Electronic Common Technical Document |
| °F | Fahrenheit |
| F | Relative bioavailability |
| FDA | Food and Drug Administration |
| $FEV_1$ | Forced Expiratory Volume (flow rate) in 1 second |
| FVC | Forced Volume Vital Capacity |
| HR | Heart Rate |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| IRB | Institutional Review Board |
| kg | Kilograms |
| mcg | Microgram |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | modified Intent-to-Treat |
| mL | Milliliter |
| NAEPP | National Asthma Education and Prevention Program |
| OGD | Office of Generic Drugs |
| $PC_{20}$ | Concentration (mg/mL) of methacholine required to reduce FEV <sub>1</sub> by 20% |
| PD | Pharmacodynamic |
| PP | Per-Protocol |
| RR | Respiratory Rate |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis Software |

**SDTM** 

Study Data Tabulation Model

| Albuterol Sulfate Inhalation Aerosol | Protocol / Study No | o. CLR | 17 | 08/ |
|---|---|---|---|---|

| T. | ABLE OF CONTENTS | |
|---|---|---|
| _] | Toc533144464 | |
| 1. | INTRODUCTION | 8 |
| | OBJECTIVES | |
| | OVERALL STUDY DESIGN | |
| 4. | IDENTITY O F INVESTIGATIONAL PRODUCT | 13 |
| 5. | RANDOMIZATION AND BLINDING. | 13 |
| | SAMPLE SIZE | |
| | STUDY POPULATIONS | |
| 8. | STATISTICAL ANALYSIS METHODS | 16 |
| | 8.1 Baseline Characteristics | |
| | 8.1.1 Patient Disposition | |
| | 8.1.2 Demographic and Other Baseline Characteristics | |
| | 8.1.3 Medical History | |
| | 8.1.4 Concomitant Medications | |
| | 8.2 Pharmacodynamic Equivalence Analyses. | |
| | 8.2.1 Primary Pharmacodynamic Endpoint | |
| | 8.2.2 Population. | |
| | 8.2.3 PC <sub>20</sub> Log Transformation | |
| | 8.2.4 NONMEM® Dataset Preparation | |
| | 8.2.5 Dose-Scale Approach | |
| | 8.2.6 Dose Response Emax Model. | |
| | 8.2.7 Alternative Approach to the Dose Response Emax Model | |
| | 8.2.8 Bootstrap | |
| | 8.2.9 Calculation of Confidence Intervals for Frel | |
| | 8.2.10 Calculation of Confidence Intervals for F <sub>rel</sub> | |
| | 8.3 Safety Analysis | |
| | 8.3.1 Adverse Events | |
| | 8.3.2 Vital Signs | |
| | 8.3.3 Physical Exam | |
| | 8.3.4 12-lead ECG | |
| | 8.3.5 Pregnancy Test | |
| | 8.3.6 Concentration of Methacholine Required to Reduce FEV <sub>1</sub> by 20% (PC <sub>20</sub> ) | |
| | 8.3.7 Forced Expiratory Volume (flow rate) in 1 second (FEV <sub>1</sub> ) | |
| | 8.3.8 Protocol Deviations | |
| | 8.4 Multiple Comparisons | |
| | 8.5 Methods for Handling Missing Data. | |
| | 8.6 Interim Analyses | |
| 9. | TABLE, LISTING AND FIGURE SHELLS | |
| | T16.1.9.1 Summary of Patient Disposition. | |
| | T16.1.9.2 Summary of Protocol Deviations. | 30 |

| 1 | ibuterol Sulfate Innalation Aerosol Protocol / Study No. CLR 1/ 08/ | |
|---|---|---|
| | T16.1.9.3 Summary of Patient's Treatments Included in the Pharmacodynamic | |
| | Analysis | 3 |
| | T16.1.9.4 Summary of Demographic Data and Baseline Characteristics | 32 |
| | T16.1.9.5 Summary of Demographic Data and Baseline Characteristics | 34 |
| | T16.1.9.6 Summary of Demographic Data and Baseline Characteristics | |
| | T16.1.9.7 Summary of Concentration (mg/mL) of Methacholine Required to Reduce | |
| | FEV <sub>1</sub> by 20% (PC <sub>20</sub> ) | 3: |
| | T16.1.9.8 Summary of Concentration (mg/mL) of Methacholine Required to Reduce | |
| | FEV <sub>1</sub> by 20% (PC <sub>20</sub> ) | 3 |
| | T16.1.9.9 Summary of Concentration (mg/mL) of Methacholine Required to Reduce | |
| | FEV <sub>1</sub> by 20% (PC <sub>20</sub> ) | 3 |
| | T16.1.9.10 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 | |
| | second (FEV <sub>1</sub> ) | 30 |
| | T16.1.9.11 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 | |
| | second (FEV <sub>1</sub> ) | 3′ |
| | T16.1.9.12 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 | |
| | second (FEV <sub>1</sub> ) | 3′ |
| | T16.1.9.13 Overall Summary of Adverse Events | |
| | T16.1.9.14.1 Summary of Frequency of All Adverse Events by System Organ Class | 39 |
| | T16.1.9.14.2 Summary of Frequency of Serious Adverse Events by System Organ | |
| | Class | 40 |
| | T16.1.9.15.1 Summary of Frequency of All Adverse Events by Relationship to Study | |
| | Drug | 4 |
| | T16.1.9.15.2 Summary of Frequency of Serious Adverse Events by Relationship to | |
| | Study Drug | 42 |
| | T16.1.9.16.1 Summary of Frequency of All Adverse Events by Severity | 43 |
| | T16.1.9.16.2 Summary of Frequency of Serious Adverse Events by Severity | |
| | T16.1.9.17 Summary of Vital Signs | 4: |
| | L16.2.1 Listing of Discontinued Subjects | 40 |
| | L16.2.2 Listing of Protocol Deviations | 4 |
| | L16.2.3.1 Listing of Subjects Excluded from the Per-Protocol Population | 48 |
| | L16.2.3.2 Listing of Subjects Excluded from the Pharmacodynamic Population | 49 |
| | L16.2.4.1 Listing of Demographic Data | |
| | L16.2.4.2 Listing of Medical History | 5 |
| | L16.2.4.3 Listing of Concomitant Medication. | 52 |
| | L16.2.5 Listing of Dosing | |
| | L16.2.6.1 Listing of Methacholine Challenge and Pulse Oximetry | |
| | L16.2.6.2 Listing of Methacholine Challenge Stages | |
| | L16.2.6.3 Listing of Spirometry Test. | 5′ |
| | L16.2.7.1 Listing of Adverse Events (Safety Population Randomization Period) | 5 |
| | L16.2.7.2 Listing of Adverse Events (Safety Population Screening Period) | |
| | L16.2.7.3 Listing of Positive Pregnancy Test Results | 60 |

| Albuterol Sulfate Inhalation Aerosol | Protocol / Study No. CLR 17 08/ | |
|---|---|---|
| L16.2.7.4 Listing of Abnormal Physical 1 | Examinations | 61 |
| L16.2.8.1 Listing of Vital Signs | | 62 |

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol CLR\_17\_08

Study No. Rev 5.0 dated 08/28/2018. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol CLR\_17\_08 (Study No. Rev 5.0 dated 08/28/2018
- The final Electronic Case Report Form (eCRF) specification for Study No.

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

#### 2. OBJECTIVES

The objectives of this study are to:

- 1. Demonstrate the pharmacodynamic equivalence of the Test formulation of albuterol sulfate inhalation aerosol, eq 90 mcg base (Sun Pharmaceuticals Industries Limited) to the marketed product PROAIR® HFA (albuterol sulfate) Inhalation Aerosol, eq 90 mcg base (Teva Respiratory, LLC) using methacholine bronchoprovocation in subjects with stable, mild asthma based on National Asthma Education and Prevention Program (NAEPP) guidelines.
- 2. Compare the safety of Test, low-dose Reference, high-dose Reference, and Placebo treatments in subjects with stable, mild asthma based on NAEPP guidelines.

#### 3. OVERALL STUDY DESIGN

This randomized, single-dose, double-blind, double-dummy, four-period, four-sequence, four-treatment, Placebo and active controlled, comparative, multiple-center, crossover-design bronchoprovocation study has been designed to evaluate the pharmacodynamic equivalence of albuterol sulfate HFA inhalation aerosol, eq 90 mcg base per inhalation (Sun Pharmaceuticals

12/21/2018

■ Sun Pharmaceuticals Industries Limited ■


#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

Industries Limited) to PROAIR® HFA (albuterol sulfate) Inhalation Aerosol, eq 90 mcg base per inhalation (Teva Respiratory, LLC) in subjects with stable, mild asthma.

Approximately 123 subjects with persistent bronchial asthma will be randomized. To qualify for inclusion in the study, subjects must be at least 18 years of age, with a documented diagnosis of mild asthma as defined by the NAEPP guidelines at least 6 months before Screening.

Randomized subjects who withdraw from the study will not be replaced.

Before any study-specific procedures are performed, all subjects will read and sign the IRB-approved informed consent form.

Eligible subjects will complete 5 clinic visits as follows:

- Visit 1: Screening (Day -14 to -1)
- Visit 2: Period 1
- Visit 3: Period 2
- Visit 4: Period 3
- Visit 5: Period 4

Clinical assessments will include  $FEV_1$  taken at each visit. If reattempts are necessary, an acceptable  $FEV_1$  is defined as the highest of three to four acceptable curves obtained at each time point. FVC and  $FEV_1/FVC$  ratio [(FEV<sub>1</sub>/FVC) x 100] will also be recorded along with  $FEV_1$  measurements at each visit.

#### **Screening**

Screening evaluations will be performed in accordance with the study calendar. Clinical assessments will include: vital sign measurement, height, weight, physical examination, urine pregnancy test (for all women of childbearing potential), 12-lead electrocardiogram (ECG), and pulse oximetry (during methacholine bronchoprovocation challenges). Chest x-ray may be performed at discretion of the Investigator. Qualifying FEV<sub>1</sub> at Screening must be  $\geq$  80% of predicted value. Once Qualifying FEV<sub>1</sub> is obtained, a sterile, saline control will be administered to the subject through a nebulizer. Spirometry will be performed following the saline administration. Post-saline FEV<sub>1</sub> should not drop more than 10% from pre-saline FEV<sub>1</sub> and should be  $\geq$  70% of predicted value. If the subject fails to meet any of these requirements, the procedures must be stopped, rescue albuterol administered, and the visit should be rescheduled. All clinical assessments except height and weight will be performed at each rescheduled visit. Subjects who fail three consecutive visits will not be eligible to participate in the study. Subjects meeting post-saline FEV<sub>1</sub> criteria will undergo methacholine bronchoprovocation challenge with

12/21/2018

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

progressively increasing concentrations to determine the subject's baseline provocation concentration of inhaled methacholine required to reduce  $FEV_1$  by 20% ( $PC_{20}$ ) relative to the post-saline value. The maximum concentration of methacholine to be administered in this step will be 8 mg/mL. Subjects who do not respond to methacholine doses at or below 8 mg/mL will not be eligible for enrollment in the study.

Once the methacholine challenge test is completed, rescue albuterol will be administered and spirometry will be performed approximately 15 minutes later until the subject's  $FEV_1$  returns to within 90% of the best post-saline  $FEV_1$  or until the Principal Investigator determines that the  $FEV_1$  has stabilized and it is safe to allow the subject to leave the site. Vital signs will also be repeated.

#### **Dosing Visits**

Eligible subjects will return for four treatment visits. The first dosing visit will occur no earlier than 24 hours and no more than 14 days after Screening procedures and the interval (washout period) between dosing visits should be at least 48 hours. At each treatment visit, the following will be performed before dosing:

- Vital sign measurement
- 12-lead electrocardiogram (ECG) as the discretion of the Investigator after the initial Screening visit
- Pulse oximetry (during methacholine bronchoprovocation challenges)
- Concomitant medication update (confirming washouts)
- Adverse Events (AE) review
- Urine pregnancy test for all women of childbearing potential

A pre-treatment evaluation will be performed. This will confirm that pre-challenge  $FEV_1$  is  $\geq$  80% of predicted and within 88 and 112% of qualifying spirometry value at Screening visit. After the first inhalation of saline control is administered, the  $FEV_1$  should not drop more than 10% compared to pre-challenge value and should be  $\geq$  70% of the predicted value. If the subject fails to meet any of these requirements, the procedures must be stopped, albuterol administered, and the visit should be rescheduled. Subjects who fail three consecutive visits should be dropped from the study.

Subsequently, review of inhaler dosing technique, priming and preparation of inhalers will be performed. The subject will receive one of the four randomized study treatments. The time of last actuation will be recorded, as well as the adequacy of inhaler technique. Approximately 15

12/21/2018

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

minutes after the last inhalation of study treatment, a methacholine bronchoprovocation challenge will be given with progressive concentrations to determine the  $PC_{20}$ . The 20% reduction in  $FEV_1$  will be determined relative to the post-saline  $FEV_1$ . After the procedures have been completed, albuterol will be administered to reverse airway obstruction and subjects will be followed until  $FEV_1$  returns to within 90% of the best  $FEV_1$  captured during the saline stage on that study day or until the Principal Investigator determines that the  $FEV_1$  has stabilized and it is safe to allow the subject to leave the site.

Subjects who withdraw prematurely will be evaluated at a final visit, but spirometry, chest x-rays, and methacholine administration do not need to be performed.

The spirometry procedures and the methacholine bronchoprovocation challenges in this study are to be performed in accordance with the ATS Guidelines for Methacholine and Exercise Challenge Testing. The maximum methacholine dose administered will be 8 mg/mL at Screening and 128 mg/mL for treatment visits.

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

Figure 1: Study Schematic

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 |
|---|---|---|---|---|---|
| Procedures | Screening | Period 1 | Period 2 | Period 3 | Period 4<br>End of Study |
| Informed Consent | X | | | | |
| Baseline Demographics | X | | | | |
| Medical History | X | | | | |
| Vital Signs* | X | X | X | X | X |
| Height and Weight | X | | | | |
| Physical Exam | X | | | | X |
| Urine Pregnancy Test** | X | X | X | X | X |
| 12-Lead ECG | X | Χ <sup>†</sup> | $X^{\dagger}$ | Χ <sup>†</sup> | Χ <sup>†</sup> |
| Chest X-Ray <sup>‡</sup> | X | | | | |
| Concomitant Medication | X | X | X | X | X |
| Spirometry (FEV <sub>1</sub> and FVC) <sup>§</sup> | X | X | X | X | X |
| Saline Control Administration | X | X | X | X | X |
| Methacholine Challenge | X | X | X | X | X |
| Pulse Oximetry | X | X | X | X | X |
| Inclusion/Exclusion Criteria<br>Review | X | | | | |
| Prime, dispense study product and instructions | | X | X | X | X |
| Dosing | | X | X | X | X |
| Assessment of Compliance | | X | X | X | X |
| Adverse Events | X | X | X | X | X |
| Provide Diary | X | X | X | X | |
| Collect /Review Diary | | X | X | X | X |
| Schedule next visit | X | X | X | X | |

<sup>\*</sup> Vital signs will be measured before and after methacholine bronchoprovocation challenges at all visits.

<sup>\*\*</sup> Female subjects of childbearing potential.

<sup>† 12-</sup>lead ECG to be performed at Screening may be repeated before methacholine bronchoprovocation challenges at discretion of Investigator.

<sup>‡</sup> Chest X-ray is to be performed at discretion of Investigator.

 $<sup>\</sup>S$  FEV $_1$  and FVC measurements will be performed before saline control, after saline control, and after methacholine administration. If reattempts are necessary, an acceptable FEV $_1$  is defined as the highest of three to four acceptable curves obtained at each time point.

<sup>|</sup> Subjects will receive four puffs of study product from four different inhalers (each dose from a separate inhaler).

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

#### 4. IDENTITY OF INVESTIGATIONAL PRODUCT

The following products will be used in the study:

**Test (T active)**: Albuterol Sulfate Inhalation Aerosol, eq 90 mcg base per inhalation (Sun Pharmaceuticals Industries Limited)

**Reference (R active)**: PROAIR® HFA (albuterol sulfate) Inhalation Aerosol, eq 90 mcg base per inhalation (Teva Respiratory, LLC)

**Test Placebo** (**T Placebo**): Placebo for Albuterol Sulfate Inhalation Aerosol (i.e., vehicle canister with T active actuator [Sun Pharmaceuticals Industries Limited])

**Reference Placebo (R Placebo)**: Placebo for Albuterol Sulfate Inhalation Aerosol (i.e., vehicle canister with R active actuator [Sun Pharmaceuticals Industries Limited])

Treatments will be as follows:

| Treatment A: Zero-dose Two different Reference Placebo inhalers and two different Test Placebo inhalers | 1 puff Inhaler 1<br>1 puff Inhaler 2<br>1 puff Inhaler 3<br>1 puff Inhaler 4 |
|---|---|
| Treatment B: 90 mcg of Reference One Reference inhaler, one Reference Placebo inhaler, and two different Test Placebo inhalers | 1 puff Inhaler 1<br>1 puff Inhaler 2<br>1 puff Inhaler 3<br>1 puff Inhaler 4 |
| Treatment C: 180 mcg of Reference Two different Reference inhalers and two different Test Placebo inhalers | 1 puff Inhaler 1<br>1 puff Inhaler 2<br>1 puff Inhaler 3<br>1 puff Inhaler 4 |
| Treatment D: 90 mcg of Test One Test inhaler, one Test Placebo inhaler, and two different Reference Placebo inhalers | 1 puff Inhaler 1<br>1 puff Inhaler 2<br>1 puff Inhaler 3<br>1 puff Inhaler 4 |

#### 5. RANDOMIZATION AND BLINDING

At Visit 1 eligible subjects will be enrolled in the study, and scheduled for Visit 2. At Visit 2, eligible subjects will be randomized to one of the four sequences as shown below. Treatments

12/21/2018

■ Sun Pharmaceuticals Industries Limited ■


#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

will be administered according to a four-treatment, four-period, four-sequence design. The randomization will be generated in blocks of four with each sequence occurring once in each block.

| Sequence | Period 1 | Period 2 | Period 3 | Period 4 |
|----------|----------|----------|----------|----------|
| 1 | A | В | С | D |
| 2 | D | С | В | A |
| 3 | С | A | D | В |
| 4 | В | D | A | С |

Subjects will be randomized to a treatment regimen in a blinded fashion by assigning randomization numbers in ascending sequential order starting with the lowest available randomization number at each site. All subjects randomized will be identified by initials, date of birth, and a unique seven-digit subject number. The first two-digits will identify the Investigator site where the subject was enrolled and the last five will correspond with the randomization number of study product 'Treatment Box' assigned to the subject. A perforated or two-part label will be attached to each of the small boxes containing individual inhalers. Both pieces of the label should include the following information: Protocol number, randomization number, space for subject's initials, statement that the study product is for Investigational Use only, space for dispensing date and the Sponsor's name. In addition all subjects will be provided with written instructions on how to use the study medication. One part of the label will remain attached to the box. The other part will be removed before dispensing and attached to the study product log.

The Investigator, staff at the study site, study monitors, and data analysis/management personnel will be blinded to the patient assignment.

#### 6. SAMPLE SIZE

The sample size estimation for this study was based on data from the study by Newhouse et al. that reported the bronchoprotective effect of inhaled salbutamol (albuterol) on methacholine  $PC_{20}FEV_1$ .

12/21/2018

■ Sun Pharmaceuticals Industries Limited ■


#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

The highest within-subject coefficient of variability (COV) value for ln-transformed  $PC_{20}$  was estimated as 0.846 from the mean ratio and SD values for the  $PC_{20}$  at the 200 and 100 mcg doses (Table 1 in reference 2). Based on this COV, 98 evaluable subjects would be required in the PD population to demonstrate pharmacodynamic equivalence (i.e., 90% confidence interval on relative bioavailability [F] is within the bioequivalence limits of 0.67 to 1.50) with 90% power for a crossover study, assuming a true ratio of F = 1.1. To allow for approximately 20% of subjects that may discontinue from the study or have major protocol violations, and therefore not qualify for the PD population, up to 123 subjects will be randomized in the study.

#### 7. STUDY POPULATIONS

#### Per-Protocol (PP) Population

The PP population will include all subjects who:

- Completed all four randomized treatment periods with an evaluable PC<sub>20</sub>FEV<sub>1</sub> in each period.
- Were compliant with study treatment dosing procedures.
- Did not use any restricted concomitant medications.
- Did not have any other significant protocol deviations.

#### Pharmacodynamic (PD) Population

The PD population used in the dose-scale analyses will include subjects who:

- Completed at least one of the four randomized treatment periods with an evaluable PC<sub>20</sub>FEV<sub>1</sub>.
- Were compliant with study treatment dosing procedures.
- Did not use any restricted concomitant medications.
- Did not have any other significant protocol deviations.

## **Safety Populations**

The Safety population will include all subjects who administered at least one actuation of any of the four investigational products (Test, Reference, Test Placebo, Reference Placebo) in any of the four randomized treatment periods.

PP and PD populations will be shortlisted upon a blinded review of the data by CRO and sponsor before database lock.

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

#### 8. STATISTICAL ANALYSIS METHODS

According to standard statistical practice, the significance threshold is set to p < 0.05 (two-tailed). Data will be summarized with respect to demographic and baseline characteristics and safety variables.

For categorical variables and non-missing data, the number and percent of each category within a parameter will be calculated. For continuous variables, statistics will include n, mean, standard deviation, median, minimum and maximum values.

All statistical analyses will be conducted using Statistical Analysis System (SAS®, version 9.4 or higher).

#### 8.1 Baseline Characteristics

#### 8.1.1 Patient Disposition

The patient disposition information will be summarized overall. The number of subjects randomized will be tabulated overall. In addition, completion status and primary reason for withdrawal will be summarized overall.

#### 8.1.2 Demographic and Other Baseline Characteristics

The following subject demographic characteristics will be summarized separately in the PP, PD and Safety populations:

- Age (years)
- Sex (male/female)
- Ethnicity (Hispanic/non-Hispanic)
- Race (White, Black/African American, Native Hawaiian or Other Pacific Islander, Asian, American Indian or Alaska Native)
- Tobacco use (yes/no)
- Number of years patient suffered from symptoms caused by asthma
- Qualifying spirometry (Visit 1, Pre- and Post-saline)
- PC<sub>20</sub> FEV<sub>1</sub> at Visit 1

12/21/2018

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

Continuous variables will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, maximum); categorical variables will be described in frequencies and percentages. Summary tables will be included.

All data will be listed by patient.

## **8.1.3 Medical History**

At Visit 1, subjects will be questioned about medical history, including acute and chronic medical history and medical history relevant to their asthma.

Medical history data will be listed by patient.

#### **8.1.4 Concomitant Medications**

On Visit 1, subjects will be asked to list their current and recent ( $\leq$  6 months) medication use. During all subsequent visits, subjects will be asked about ongoing and new concomitant medications.

All prior and concomitant medications will be listed by patient.

## 8.2 Pharmacodynamic Equivalence Analyses

Pharmacodynamic (PD) equivalence between Test and Reference will be based on the dose-scale method of analysis of the post-dose  $PC_{20}$  (mg/mL) data using non-linear  $E_{max}$  modeling, as outlined in the FDA Draft Guidance on Orlistat capsule (3). Alternative models may be tested if warranted by the data, and these models as well as the specific criteria related to their use, are described in more detail in Section 8.2.7.

#### 8.2.1 Primary Pharmacodynamic Endpoint

The primary pharmacodynamic endpoint is the post-dose  $PC_{20}$ , which is the provocative concentration of methacholine challenge agent required to reduce the forced expiry volume in one second (FEV<sub>1</sub>) by 20%, following the administration of different doses of albuterol (or placebo) by inhalation.

The 20% reduction in FEV<sub>1</sub> will be determined relative to the post-saline FEV<sub>1</sub> measure before placebo or albuterol administration. The methacholine  $PC_{20}$  will be calculated by linear interpolation from the observed data relating the % decrease in  $FEV_1$  from the post-saline  $FEV_1$  to the concentration of methacholine that provokes at least a 20% decrease in  $FEV_1$ . This interpolation will be based on log transformed methacholine concentrations. In the event that subjects receiving the maximum concentration of methacholine (128 mg/mL) at any dosing visit (Visits 2-5) do not achieve at least a 20% fall in  $FEV_1$ , then they will have their  $PC_{20}FEV_1$  data recorded as > 128 mg/mL and the data from that visit will be excluded from the statistical analysis; the data from the other Visits for these subjects will be eligible for inclusion in the PD

12/21/2018

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

population but will be excluded from the PP population.

#### 8.2.2 Population

The primary dose-scale analysis will be performed using the PD population as NONMEM allows for the use of all available data, without biasing the F estimation. For information purposes only, an additional dose-scale analysis will be performed using the PP population.

### 8.2.3 PC<sub>20</sub> Log Transformation

The FDA product-specific guidance for albuterol sulfate explains that "log transformation of the PD data before fitting the Emax model is recommended for dose-scale analysis" (4); however, this guidance does not specify which log transformation should be used. Therefore, the PC<sub>20</sub> values will be transformed using the reported Log<sub>2</sub> method (5,6), prior to NONMEM® dataset construction.

The datasets will include individual albuterol dosing information and  $PC_{20}$  data. The actual dosing amount per treatment period will be used. Formulation will also be entered in the dataset. These will be entered as 0 for the reference product and 1 for the test product. The placebo dose will also be considered as the reference formulation. The dose amount for the placebo treatment will be set to 0. Data will be excluded from the analysis if insufficient or inaccurate dosing information are recorded.

#### 8.2.5 Dose-Scale Approach

To assess bioequivalence using PD endpoints, the FDA albuterol-specific guidance (4) recommends using the dose-scale approach described in FDA's orlistat guidance (3). This approach involves fitting dose-response data using the following equation:

Equation 1 Response = 
$$E_0 + \frac{E \max \cdot Dose \cdot F_{rel}}{ED_{50} + Dose \cdot F_{rel}}$$

In Equation 1, the response is the measured  $PC_{20}$ ,  $E_0$  is the baseline response, Emax is the maximal response,  $ED_{50}$  is the dose associated with half of the maximal response and  $F_{rel}$  is the relative bioavailability of the test product compared to that of the reference product. This model is based on the assumption that  $E_0$ ,  $ED_{50}$  and Emax are the same for the test and reference products.

The FDA orlistat guidance allows for the dose-scale Emax model to be fitted either to the mean or to the individual scores of dose response data. The analysis described in this plan will be

12/21/2018

■ Sun Pharmaceuticals Industries Limited ■


## Albuterol Sulfate Inhalation Aerosol Protocol / Study No. CLR 17 08/

based on each individual score because this method is generally considered more robust in a bioequivalence (BE) crossover trial.

The PC<sub>20</sub> data will be analyzed based on a two-step dose-scale analysis to estimate F<sub>rel</sub>:

- Firstly, a dose-response relationship will be mathematically described by fitting the relevant Emax model to the individual dose-response data, and an estimate for F<sub>rel</sub> will be obtained.
- Secondly, a 90% confidence interval for F<sub>rel</sub> will be estimated by using Efron's (7) biascorrected and accelerated (BCa) method.

#### 8.2.6 Dose Response Emax Model

The analysis will use the FDA recommended Emax model using NONMEM®. The model will include the following:

- Etas will be included on PD parameters  $E_0$ , Emax and  $ED_{50}$ , coded as Theta(x)+Eta(x) for  $E_0$  and Emax and as Theta(x)\*exp(Eta(x)) for  $ED_{50}$ .
- The possibility of adding an eta on the F<sub>rel</sub> parameter will be tested..
- A combination of proportional and additive residual error (Epsilons).

Additionally, the model may be simplified by removing certain parameters (Etas or Epsilons) if they are estimated to be close to the boundary (e.g., 0).

Quality of fit and selection of an alternate model will be determined using the objective function. A lower objective function is preferred if a model has the same number of parameters. Otherwise, the model will be chosen according to the difference in the MOF based on a Chisquare distribution (p < 0.01 will be considered significant), taking the difference in the numbers of fitted parameters into account. Throughout the modeling process, the first-order conditional estimate (FOCE) option in NONMEM will be used.

#### 8.2.7 Alternative Approach to the Dose Response Emax Model

The Emax model (as described in Sections 8.2.5 and 8.2.6) is the model described by the FDA in the Orlistat guidance (3) and is the preferred one. However, based on the results of this Emax model, further analysis may be required. More specifically, an alternate approach will be used to re-analyze the data if the following 2 criteria are met:

- If the predicted response of the low-dose and high-dose of albuterol fall within 20-80% of the maximum response.
- If the predicted response for the low-dose of albuterol is  $\geq 75\%$  of the predicted response for the high-dose albuterol.

12/21/2018

■ Sun Pharmaceuticals Industries Limited ■


#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

Therefore, if the Emax model previously described in this section is appropriate at describing the  $PC_{20}$  data, it will be used and will be considered final. However, if this Emax model is considered inappropriate (based on criteria listed above), the alternative modeling approach will be used as described below.

The relationship between dose and response can often be described by a hyperbolic curve that is defined by the following equation, often called the "Emax model":

Equation 2 
$$Response = \frac{Emax \cdot Dose}{Dose + D_{50}}$$

This relationship is depicted below, in Figure 1.

Figure 1. Example of Emax Dose-Response Relationship



In theory, a minimum of two observations are required to estimate the two model parameters (Emax and  $D_{50}$ ). Ideally, these two data points should be as far apart as possible, and lie close to the inflection points on the curve, to properly characterize Emax and  $D_{50}$ . This ideal scenario is depicted in Figure 2; with the predicted Emax curve in black, observed data represented by red circles, and their associated error shown by vertical lines passing through the circle's center.

Figure 2. Example of Emax Relationship with Data Points that are Spread Out



Figure 2 depicts the ideal scenario; however, in practice the data points may not always lie this far apart. If these two data points are too close to one and other, Emax and  $ED_{50}$  estimations can be more difficult and less certain.

In other words, different Emax relationships, or combinations of parameter estimates (Emax and  $ED_{50}$ ), could explain the same data points; therefore, it becomes more difficult to know with certainty which relationship reflects reality. This problem is illustrated in Figure 3, where very different Emax curves (denoted by the black, blue and yellow lines) all pass through the same two observed data points (red points with vertical error bars).

Figure 3. Example of Possible Emax Curves for the Same Data Points



If the response data associated with the two doses (90 mg and 180 mg) are close to one and other, which is analogous to the scenario depicted in Figure 3, this proximity of the data will make it difficult to properly estimate the parameters Emax and  $ED_{50}$ .

In such cases, log-transformation of the independent variable (dose) can be beneficial. The  $\log_{10}$  transformation of dose is used in such analyses. Despite the hyperbolic nature of the Emax curve, it is recognized that when the data on the X-axis are log-transformed, the relationship becomes more linear, especially between doses that are associated with 20% and 80% of Emax. (8); this is illustrated in Figure 4.

Figure 4. Depiction of Log-Linear Dose-Response Relationship



When using a log-linear model, the relationship between log(dose) and response can be described by a straight-line between 20% and 80% of the maximum effect. Consequently, it is no longer necessary to estimate Emax and  $ED_{50}$  parameters, thereby removing the uncertainty associated with these parameter estimates. Instead, the relationship between log(dose) and response can be described by a simple slope and intercept.

It can also be appreciated from Figure 4 that when using the log-linear model, the intercept (the hypothetical response at dose zero based on a linear relationship) is not equivalent to the  $E_0$  that is associated with the Emax model. Therefore, response data associated with the placebo should not be fitted by the log-linear model for two reasons:

- 1) Linearity only applies to doses that are associated with responses that are between 20% and 80% of the maximal response. By definition, this excludes a dose of zero that is not associated with a response.
- 2) Inclusion of placebo data would falsely bias the estimation of the intercept parameter, and the slope that would be fitted by the model would not reflect the true slope. Other parameter estimates (such as  $F_{rel}$ ) will also be unreliable.

For the reasons above, the placebo data should not be fitted in the log-linear model. In such an analysis, only response data associated with the 90 mg and 180 mg should be fitted by this type of model. An additional analysis may be done for which the response data associated with the 90 mg and 180 mg may be placebo-corrected to account for the placebo effect.

12/21/2018

■ Sun Pharmaceuticals Industries Limited ■


#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

Therefore, in this alternate model, PC<sub>20</sub> would be fitted according to the following equation:

Equation 3 
$$Response = Intercept + Slope * Dose * F_{rel}$$

In this relationship, both response and dose are log-transformed.

The analysis using the Emax model detailed in the previous section will be presented for information purposes only even if this alternative approach is used.

#### 8.2.8 Bootstrap

In the FDA orlistat guidance (3), 90% CI are constructed using a nonparametric bootstrap technique. Essentially, subjects are repeatedly sampled at random with replacement, creating new datasets of the same size as the original dataset and new PD parameters are estimated using the same final model. Ten thousand (10 000) of these bootstrap samples will be constructed and NONMEM<sup>®</sup> analyses will be performed on all. A matrix of bootstrap mean population estimates ( $F_{rel}$ ) will thus be obtained (9). Only the bootstrap for successful NONMEM<sup>®</sup> analyses will be used to build the 90% CI.

Bootstrapping analyses will be conducted using Wings for NONMEM® version WFN7.

#### 8.2.9 Calculation of Confidence Intervals for Frel

The bias-corrected and accelerated (BCa) method for constructing the 90% CI for  $F_{rel}$  will be employed as described in the FDA guidance for orlistat (3), using the formulae described by Efron & Tibshirani (7).

The BCa interval of intended coverage 1-2 $\alpha$  is given by Equation 4, where  $\hat{\theta}^{*(\alpha_1)}$  and  $\hat{\theta}^{*(\alpha_2)}$  are the  $100 \cdot \alpha_1^{th}$  and  $100 \cdot \alpha_2^{th}$  percentiles of the B bootstrap replications, respectively. The variables  $\alpha_1$  and  $\alpha_2$  are defined in Equations 5a and 5b.

Equation 4 
$$BC_a: (\hat{\theta}^{*(\alpha_1)}, \hat{\theta}^{*(\alpha_2)})$$

Equations 5a 
$$\alpha_1 = \Phi \left( \hat{z}_0 + \frac{\hat{z}_0 + z^{(\alpha)}}{1 - \hat{a} \cdot (\hat{z}_0 + z^{(\alpha)})} \right)$$

Equation 5b 
$$\alpha_2 = \Phi \left( \hat{z}_0 + \frac{\hat{z}_0 + z^{(1-\alpha)}}{1 - \hat{a} \cdot (\hat{z}_0 + z^{(1-\alpha)})} \right)$$

12/21/2018

■ Sun Pharmaceuticals Industries Limited ■


#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

In Equations 5a and 5b,  $\Phi(\cdot)$  represents the standard normal cumulative distribution function and  $z^{(\alpha)}$  is the  $100 \cdot \alpha^{th}$  percentile point of a standard normal distribution. The variables  $\hat{a}$  and  $\hat{z}_0$  represent acceleration and bias-correction, respectively. They are computed as described by Equations 6 and 7.

Equation 6 
$$\hat{z}_0 = \Phi^{-1} \left( \frac{\# \left\{ \hat{\theta}^*(b) < \hat{\theta} \right\}}{B} \right)$$

Equation 7 
$$\hat{a} = \frac{\sum_{i=1}^{n} (\hat{\theta}_{(\cdot)} - \hat{\theta}_{(i)})^{3}}{6 \left[ \sum_{i=1}^{n} (\hat{\theta}_{(\cdot)} - \hat{\theta}_{(i)})^{2} \right]^{3/2}}$$

In Equation 6,  $\Phi^{-1}(\cdot)$  indicates the inverse function of a standard normal cumulative distribution function. The numerator represents the number of bootstrap values  $\hat{\theta}^*(b)$  that are less than the original estimate of  $\hat{\theta}$ . B is the number of bootstrap replicates.

Equation 7 uses  $\hat{\theta}_{(i)}$  and  $\hat{\theta}_{(i)}$ , which are the average values of all jackknife replications and the i<sup>th</sup> jackknife replication of  $\hat{\theta}$ , respectively.

The calculation of the BCa interval will be performed with the code provided by Efron & Tibshirani (10), using S-Plus for Windows<sup>®</sup>.

#### 8.2.10 Calculation of Confidence Intervals for F<sub>rel</sub>

The test formulation will be declared bioequivalent to the reference formulation if the estimated  $F_{rel}$  and the 90% CI are completely contained within the range of 67.00 to 150.00%.

### 8.3 Safety Analysis

All study subjects who administered at least one actuation of any of the study products (Safety Population) will be included in the comparative safety analysis.

#### 8.3.1 Adverse Events

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary

12/21/2018

■ Sun Pharmaceuticals Industries Limited ■


#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

(Version 20.0 or higher). Each adverse event is to be evaluated for date of start and end, seriousness, severity, causal relationship with the study drugs, action taken and outcome.

A summary table of the number and percent of subjects with AEs by system organ class, preferred term, will be presented. Each patient will be counted only once within each preferred term. Other summaries may be added based on the data obtained.

A frequency summary table of the number of AEs by system organ class, preferred term, and severity will be presented. Severity will be classified as "Mild", "Moderate" or "Severe".

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to a study drug will be presented. Relationship to a study drug will be classified as "Not Related" or "Related" where causality "Certain, Probable and Possible" will be assessed as "Related" while "Unlikely and Unrelated" will be assessed as "Not Related".

A frequency summary table of the number of SAEs by system organ class, preferred term will also be presented by treatment group.

If sufficient data exist, AEs frequencies will be compared among treatments using Fisher's exact test. If the overall Fisher's exact test is significant for comparisons across the 4 treatments, pairwise testing between treatments will be conducted to determine which contrasts are significant.

All AEs will be listed by patient for the Safety Population.

#### 8.3.2 Vital Signs

At each clinic visit, subjects' vital signs (pulse, BP, temperature, and respiration rate) will be recorded before and after methacholine procedures.

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided by treatment and time point.

All data will be listed by patient.

#### 8.3.3 Physical Exam

At Visits 1 and 5, the Investigator will perform a general physical exam for each qualified patient; any significant findings will be noted. At minimum, the physical exam must include a head, ear, eyes, nose, lungs and throat examination.

Any abnormal physical exam results will be listed by patient and visit.

#### 8.3.4 12-lead ECG

Subjects will undergo a 12-lead ECG at Screening. An ECG may be performed at subsequent visits at the Investigator's discretion. Any clinically significant findings will be noted.

12/21/2018

■ Sun Pharmaceuticals Industries Limited ■


#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. CLR 17 08/

12-lead ECG results will be listed by patient and visit.

### 8.3.5 Pregnancy Test

Urine pregnancy tests on women of childbearing potential will be performed at each clinic visit, including rescheduled visits.

Positive urine pregnancy test results will be listed by patient and visit.

#### 8.3.6 Concentration of Methacholine Required to Reduce FEV<sub>1</sub> by 20% (PC<sub>20</sub>)

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided separately for  $PC_{20}$  by treatment for the PP, PD and Safety Population.

### 8.3.7 Forced Expiratory Volume (flow rate) in 1 second (FEV<sub>1</sub>)

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided separately for pre-challenge FEV<sub>1</sub> by visit for the PP, PD and Safety Population.

#### 8.3.8 Protocol Deviations

The total number of subjects with protocol deviation, the total number of protocol deviations as well as protocol deviation categories will be summarized.

Protocol deviations will be listed by patient.

#### **8.4 Multiple Comparisons**

No multiple comparison adjustment will be made in this study.

#### 8.5 Methods for Handling Missing Data

Each demographic and baseline characteristic variable will be analyzed using all available data. Thus, subjects with missing data will only be excluded from analyses for which data are not available.

#### 8.6 Interim Analyses

No interim analyses are planned for this study.

#### 9. TABLE, LISTING AND FIGURE SHELLS

The following shells are included to provide a framework for displaying data in the final clinical study report. These shells are meant to provide a general layout for final Tables, Listings and Figures; therefore, they may not reflect every aspect of the current study.

Tables, Listings and Figures are numbered in accordance with the ICH structure. Following data

12/21/2018

■ Sun Pharmaceuticals Industries Limited ■


## Albuterol Sulfate Inhalation Aerosol

Protocol / Study No. CLR 17 08/

analyses, table headers, variables names and footnotes will be modified as needed.

Descriptive and inferential statistical (including bootstrap) analyses will be performed using SAS® statistical software version 9.4 or higher and NONMEM®, unless otherwise noted.

**T16.1.9.1 Summary of Patient Disposition** 

| Subjects | Overall<br>(n (%)) |
|---------------------|--------------------|
| Subjects Screened | XX |
| Subjects Randomized | XX |
| Safety Population | XX |
| Completed Study | xx (xx.x) |
| Terminated Early | xx (xx.x) |
| Adverse Event | xx (xx.x) |
| Lack of Efficacy | xx (xx.x) |
| Lost to follow-up | xx (xx.x) |
| etc. | xx (xx.x) |
| | xx (xx.x) |
| Other | xx (xx.x) |

<sup>%</sup> is based on total number of subjects in the safety population.

Created on: ddmmmyy hh:mm

Page 1 of N

# T16.1.9.2 Summary of Protocol Deviations (Safety Population)

| | Total<br>N = xx |
|-----------------------------------------|-----------------|
| Total Subjects with Protocol Deviations | XX |
| Total Deviations | XX |
| Assessment conducted out of window | XX |
| Lost to Follow-up | XX |
| Missed Visit | XX |
| Non-compliance with study drug | XX |
| Non-compliance with study procedures | XX |
| Restricted Medication | XX |
| etc. | XX |
| | XX |
| Other | XX |

Created on: ddmmmyy hh:mm Page 1 of N

## **Albuterol Sulfate Inhalation Aerosol**

## Protocol / Study No. AI CLR 17 08/

## T16.1.9.3 Summary of Patient's Treatments Included in the Pharmacodynamic Analysis

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Treatment A | Treatment B | Treatment C | Treatment D |
|---|---|---|---|---|---|---|
| XX-XXXX | xx-xxxxx | 1 | Yes | Yes | Yes | No |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

Created on: ddmmmyy hh:mm Page 1 of N

T16.1.9.4 Summary of Demographic Data and Baseline Characteristics (Safety Population)

| | | $ \begin{array}{l} \text{Total} \\ \text{N} = xx \end{array} $ |
|---|---|---|
| Age (years) | n | XX |
| | Mean $\pm$ SD | $xx.x \pm x.x$ |
| | Median | XX.X |
| | Range | XX-XX |
| Race (n (%)) | American Indian or Alaska Native | xx (xx.x) |
| | Asian | xx (xx.x) |
| | Black/African American | xx (xx.x) |
| | Native Hawaiian or other Pacific Islander | xx (xx.x) |
| | White | xx (xx.x) |
| | Other | xx (xx.x) |
| Ethnicity (n (%)) | Hispanic or Latino | xx (xx.x) |
| | Not Hispanic or Latino | xx (xx.x) |
| Gender (n (%)) | Female | xx (xx.x) |
| | Male | xx (xx.x) |
| Tobacco use (n (%)) | Yes | xx (xx.x) |
| | No | xx (xx.x) |
| Number of years patient has suffered from symptoms caused by asthma | n | XX |
| | $Mean \pm SD$ | $xx.x \pm x.x$ |
| | Median | XX.X |
| | Range | xx-xx |
#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

| | | Total N = xx |
|-----------------------------------|---------------|----------------|
| FEV <sub>1</sub> (L) (Pre-saline) | n | XX |
| | $Mean \pm SD$ | $xx.x \pm x.x$ |
| | Median | XX.X |
| | Range | XX-XX |
| $FEV_1(L)$ (Post-saline) | n | XX |
| | $Mean \pm SD$ | $xx.x \pm x.x$ |
| | Median | XX.X |
| | Range | XX-XX |
| $PC_{20} FEV_1 $ (mg/mL) | n | XX |
| | $Mean \pm SD$ | $xx.x \pm x.x$ |
| | Median | XX.X |
| | Range | XX-XX |

N= number of subjects in the safety population; n= number of subjects with data available; % is based on N

Created on: ddmmmyy hh:mm

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. AI CLR 17 08/

Similar table will be created for:

T16.1.9.5 Summary of Demographic Data and Baseline Characteristics (Pharmacodynamic Population)

T16.1.9.6 Summary of Demographic Data and Baseline Characteristics (Per-Protocol Population)

T16.1.9.7 Summary of Concentration (mg/mL) of Methacholine Required to Reduce FEV<sub>1</sub> by 20% (PC<sub>20</sub>) (Safety Population)

| Statistic | Treatment A N = xx | Treatment B N = xx | Treatment C<br>N = xx | Treatment D<br>N = xx |
|---|---|---|---|---|
| n | XX | XX | XX | XX |
| Mean $\pm$ SD | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ |
| Median | XXX.X | XXX.X | XXX.X | XXX.X |
| Range | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |

Created on: ddmmmyy hh:mm Page 1 of N

T16.1.9.8 Summary of Concentration (mg/mL) of Methacholine Required to Reduce FEV<sub>1</sub> by 20% (PC<sub>20</sub>) (Pharmacodynamic Population)

T16.1.9.9 Summary of Concentration (mg/mL) of Methacholine Required to Reduce  $FEV_1$  by 20% (PC<sub>20</sub>) (Per-Protocol Population)

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. AI CLR 17 08/

T16.1.9.10 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 second (FEV<sub>1</sub>) (Safety Population)

| Visit | Statistic | Overall |
|-----------------------|---------------|------------------|
| Visit 1 (Pre-saline) | N | XX |
| | Mean $\pm$ SD | $xxx.x \pm xx.x$ |
| | Median | XXX.X |
| | Range | xxx.x - xxx.x |
| Visit 1 (Post-saline) | N | XX |
| | Mean $\pm$ SD | $xxx.x \pm xx.x$ |
| | Median | XXX.X |
| | Range | xxx.x - xxx.x |
| Visit 2 (Pre-saline) | N | XX |
| | Mean $\pm$ SD | $xxx.x \pm xx.x$ |
| | Median | XXX.X |
| | Range | xxx.x - xxx.x |
| Visit 2 (Post-saline) | N | XX |
| , , , | Mean $\pm$ SD | $xxx.x \pm xx.x$ |
| | Median | XXX.X |
| | Range | xxx.x - xxx.x |
| Visit 3 (Pre-saline) | · · | |
| Visit 3 (Post-saline) | | |
| Visit 4 (Pre-saline) | | |
| Visit 4 (Post-saline) | | |
| Visit 5 (Pre-saline) | | |
| Visit 5 (Post-saline) | | |

Created on: ddmmmyy hh:mm

Protocol / Study No. AI CLR 17 08/

T16.1.9.11 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 second (FEV<sub>1</sub>) (Pharmacodynamic Population)

T16.1.9.12 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 second (FEV<sub>1</sub>)

(Per-Protocol Population)

T16.1.9.13 Overall Summary of Adverse Events (Safety Population)

| Description | Treatment A N = xx n (%) | Treatment B N = xx n (%) | Treatment C N = xx n (%) | Treatment D N = xx n (%) | Total<br>N = xx<br>n (%) |
|---|---|---|---|---|---|
| Subjects in Safety Analysis Population | XX | XX | XX | XX | XX |
| Subjects with at least one AE | xx (xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Discontinued study drug due to above AEs | xx(xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| AEs reported | XX | XX | XX | XX | XX |
| Mild | xx (xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Moderate | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| Severe | xx (xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Not Related | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| Related | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| Serious AE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) |

<sup>&</sup>quot;Certain, Probable and Possible" were assessed as "Related" while "Unlikely and Unrelated" were assessed as "Not Related".

Created on: ddmmmyy hh:mm

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. AI CLR 17 08/

T16.1.9.14.1 Summary of Frequency of All Adverse Events by System Organ Class (Safety Population)

| | Treatment A $N = xx$ | | Treatment B N = xx | | | Treatment C<br>N = xx | | Treatment D<br>N = xx | |
|---|---|---|---|---|---|---|---|---|---|
| Body System/<br>MedDRA Term | Events | Subjects<br>n (%) | Events | Subjects<br>n (%) | Events | Subjects<br>n (%) | Events | Subjects<br>n (%) | Fisher's<br>P-value |
| Patient with at least one AE | XX | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | XX | xx (xx.x) | X.XXXX |
| Ear and labyrinth disorders/ Ear pain | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | X.XXXX |

etc.

N= number of subjects in the safety population in that particular group; n= number of subjects with data available for that particular group; % is based on N

**Programming Note**: Note that if the overall Fisher's exact test is significant for comparisons across the 4 treatments then pair-wise testing between treatments will be conducted to determine which contrasts are significant.

Created on: ddmmmyy hh:mm

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. AI CLR 17 08/

T16.1.9.14.2 Summary of Frequency of Serious Adverse Events by System Organ Class (Safety Population)

| | Treatment A N = xx | | Treatment B<br>N = xx | | Treatment C<br>N = xx | | Treatment D<br>N = xx | | |
|---|---|---|---|---|---|---|---|---|---|
| Body System/<br>MedDRA Term | Events | Subjects<br>n (%) | Events | Subjects<br>n (%) | Events | Subjects<br>n (%) | Events | Subjects<br>n (%) | Fisher's<br>P-value |
| Patient with at least one AE | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | X.XXXX |
| Ear and labyrinth disorders/ Ear pain | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | X.XXXX |

etc.

N= number of subjects in the safety population in that particular group; n= number of subjects with data available for that particular group; % is based on N

**Programming Note**: Note that if the overall Fisher's exact test is significant for comparisons across the 4 treatments then pair-wise testing between treatments will be conducted to determine which contrasts are significant.

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. AI CLR 17 08/

T16.1.9.15.1 Summary of Frequency of All Adverse Events by Relationship to Study Drug (Safety Population)

| | Treatment A N = xx | | Treatment B $N = xx$ | | | ment C<br>= xx | Treatment D $N = xx$ | |
|---|---|---|---|---|---|---|---|---|
| Body System/<br>MedDRA Term | Related n (%) | Not<br>Related<br>n (%) | Related<br>n (%) | Not<br>Related<br>n (%) | Related<br>n (%) | Not Related<br>n (%) | Related n (%) | Not Related<br>n (%) |
| Patient with at least one AE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ear and labyrinth disorders/ Ear pain | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N= number of subjects in the safety population in that particular group; n= number of subjects with data available for that particular group; % is based on N

Created on: ddmmmyy hh:mm

<sup>&</sup>quot;Certain, Probable and Possible" were assessed as "Related" while "Unlikely and Unrelated" were assessed as "Not Related".

T16.1.9.15.2 Summary of Frequency of Serious Adverse Events by Relationship to Study Drug (Safety Population)

| | Treatment A N = xx | | Treatment B $N = xx$ | | | ment C<br>= xx | Treatment D $N = xx$ | |
|---|---|---|---|---|---|---|---|---|
| Body System/<br>MedDRA Term | Related n (%) | Not<br>Related<br>n (%) | Related n (%) | Not<br>Related<br>n (%) | Related<br>n (%) | Not Related<br>n (%) | Related n (%) | Not Related<br>n (%) |
| Patient with at least one AE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ear and labyrinth disorders/ Ear pain | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N= number of subjects in the safety population in that particular group; n= number of subjects with data available for that particular group; % is based on N

Created on: ddmmmyy hh:mm

<sup>&</sup>quot;Certain, Probable and Possible" were assessed as "Related" while "Unlikely and Unrelated" were assessed as "Not Related".

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. AI CLR 17 08/

T16.1.9.16.1 Summary of Frequency of All Adverse Events by Severity (Safety Population)

| | _ | atment A | | Treatment B N = xx | | | Treatment C $N = xx$ | | | Treatment D $N = xx$ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Body System/<br>MedDRA Term | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) |
| Patient with at least one AE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ear and labyrinth disorders/ Ear pain | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N= number of subjects in the safety population in that particular group; n= number of subjects with data available for that particular group; % is based on N

Created on: ddmmmyy hh:mm

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. AI CLR 17 08/

T16.1.9.16.2 Summary of Frequency of Serious Adverse Events by Severity (Safety Population)

| | _ | eatment A<br>N = xx | | Treatment B N = xx | | | Treatment C<br>N = xx | | | Treatment D $N = xx$ | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Body System/<br>MedDRA Term | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) |
| Patient with at least one AE | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ear and labyrinth disorders/ Ear pain | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N= number of subjects in the safety population in that particular group; n= number of subjects with data available for that particular group; % is based on N

Created on: ddmmmyy hh:mm

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. AI CLR 17 08/

# T16.1.9.17 Summary of Vital Signs (Safety Population)

| Vital Signs | Time<br>Point | Statistic | Treatment A N = xx | Treatment B $N = xx$ | Treatment C<br>N = xx | Treatment D<br>N = xx |
|---|---|---|---|---|---|---|
| Systolic Blood Pressure (mmHg) | Pre-Challenge | n | Xx | XX | XX | XX |
| | | $Mean \pm SD$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ |
| | | Median<br>Range | $\begin{array}{c} xxx.x \\ xxx.x - xxx.x \end{array}$ | $\begin{array}{c} xxx.x \\ xxx.x - xxx.x \end{array}$ | xxx.x $xxx.x - xxx.x$ | $\begin{array}{c} xxx.x \\ xxx.x - xxx.x \end{array}$ |
| | Post-Challenge | _ | | | | |

Diastolic Blood Pressure (mmHg) Pulse Rate (beats/min) Respiration Rate (breaths/min) Temperature (F)

Created on: ddmmmyy hh:mm

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.1 Listing of Discontinued Subjects

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Date of<br>Early Termination | Early Termination<br>Reason |
|---|---|---|---|---|
| XX-XXXX | XX-XXXXX | 1 | yyyy-mm-dd | Lost to Follow-up |

G 1 A DOD A DODA A GADD A DDAG

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# **L16.2.2 Listing of Protocol Deviations**

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Event Description |
|---|---|---|---|
| XX-XXXX | XX-XXXXX | 1 | Outside Visit Window (Visit 3) |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.3.1 Listing of Subjects Excluded from the Per-Protocol Population

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Exclusion Reason |
|---|---|---|---|
| XX-XXXX | XX-XXXXX | 1 | Patient did not meet IE criterion |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.3.2 Listing of Subjects Excluded from the Pharmacodynamic Population

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Exclusion Reason |
|---|---|---|---|
| xx-xxxx | XX-XXXXX | 1 | Patient did not meet IF criterion |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.4.1 Listing of Demographic Data

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Age<br>(yrs) | Gender | Ethnicity | Race |
|---|---|---|---|---|---|---|
| XX-XXXX | XX-XXXXX | 1 | 21 | Female | Not Hispanic or Latino | Black or African American |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.4.2 Listing of Medical History

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | System | Diagnosis or<br>Surgical<br>Procedure | Start Date | End Date | Ongoing |
|---|---|---|---|---|---|---|---|
| XX-XXXX | xx-xxxxx | 1 | xxxxxxxxxxxx | xxxxxxxxxx | yyyy-mm-dd | yyyy-mm-dd | |
| xx-xxxx | xx-xxxx | 2 | xxxxxxxxxxxxx | Xxxxxxxxxx | yyyy-mm-dd | | Ongoing |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

#### Protocol / Study No. AI CLR 17 08/

# L16.2.4.3 Listing of Concomitant Medication

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Medication | Dosage | Frequency* | Route | Start/End<br>Date | Indication |
|---|---|---|---|---|---|---|---|---|
| XX-XXXX | xx-xxxxx | 1 | Lisinopril | 20 MG | QD | PO | yyyy-mm-dd /<br>yyyy-mm-dd | Hypertension |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

\*PRN - As needed; QD - Daily (once per day); Q4H - Every 4 hours; Q8H - Every 8 hours; Q12H - Every 12 hours; BID - Twice per day; TID - 3 times per day; QID - 4 times per day; QOD - Every other day; QS - Every week; QM - Every month; Q3M - Every 3 months

Created on: ddmmmyy hh:mm

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.5 Listing of Dosing

| Patient<br>Screen<br>Number | Patient<br>Randomi<br>zation<br>Number | Sequence | Visit | Is the<br>Patient<br>Eligible for<br>Dosing? | First<br>Actuation<br>Time | Last<br>Actuation<br>Time | Was the Study<br>Product<br>Primed? | Was the Patient<br>Instructed on<br>How to Properly<br>Dose? | Dispenser Observe<br>the Study<br>Product Was<br>Administered? | Was the Patient<br>Compliant with the<br>Dosing Instruction? |
|---|---|---|---|---|---|---|---|---|---|---|
| xx-xxxx | xx-xxxxx | 1 | Visit 2 | Yes | hh:mm | hh:mm | Yes | Yes | Yes | Yes |
| | | | Visit 3 | Yes | hh:mm | hh:mm | Yes | Yes | Yes | No (Spray mist was seen) |
| | | | Visit 4 | Yes | hh:mm | hh:mm | Yes | Yes | Yes | Yes |
| | | | Visit 5 | Yes | hh:mm | hh:mm | Yes | Yes | Yes | Yes |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.6.1 Listing of Methacholine Challenge and Pulse Oximetry

| Patient<br>Screen<br>Number | Patient<br>Randomi-<br>zation<br>Number | Sequence | Visit | Methacholine<br>Bronchoprovocation<br>Challenge<br>Administration Time | Time FEV <sub>1</sub> Reduced by $\geq 20\%$ | Treatment<br>Dose (mcg) | PC <sub>20</sub> (mg/mL) | Pulse<br>Oximetry<br>Time | Pulse<br>Oximetry<br>(%) | FEV <sub>1</sub> at Time<br>of Discharge<br>(L) |
|---|---|---|---|---|---|---|---|---|---|---|
| XX-XXXX | XX-XXXXX | 1 | Visit 1 | hh:mm | hh:mm | NA | XXX.X | hh:mm | XX.X | xxx.x |
| | | | Visit 2 | hh:mm | hh:mm | Placebo, 0 | xxx.x | hh:mm | XX.X | XXX.X |
| | | | Visit 3 | hh:mm | hh:mm | Test, 90 | XXX.X | hh:mm | XX.X | xxx.x |
| | | | Visit 4 | hh:mm | hh:mm | Reference, 90 | XXX.X | hh:mm | XX.X | xxx.x |
| | | | Visit 5 | hh:mm | hh:mm | Reference, 180 | XXX.X | hh:mm | XX.X | XXX.X |

Note: Methacholine Bronchoprovocation Challenge administration time refers to the time of the start of the first MC bronchoprovocation challenge administration.

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. AI CLR 17 08/

L16.2.6.2 Listing of Methacholine Challenge Stages

| Patient<br>Screen<br>Number | Patient<br>Randomi-<br>zation<br>Number | Sequence | Visit | StageN | Stage | FEV <sub>1</sub> | FVC | FEV <sub>1</sub> /FVC x 100 |
|---|---|---|---|---|---|---|---|---|
| xx-xxxx | xx-xxxxx | 1 | Visit 1 | -1 | Pre-Saline | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 1 | 0 | Post-Saline | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 1 | 1 | 0.0312 | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 1 | 2 | 0.0625 | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 1 | 3 | 0.1250 | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 1 | 4 | 0.2500 | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 1 | 5 | 0.5000 | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 1 | 6 | 1.0000 | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 1 | 7 | 2.0000 | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 1 | 8 | 4.0000 | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 1 | 9 | 8.0000 | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 1 | 10 | Recovery | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 2 | -1 | Pre-Saline | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 2 | 0 | Post-Saline | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 2 | 1 | 0.0312 | X.XXX | x.xxx | XX.XXXX |
| | | | Visit 2 | 2 | 0.0625 | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 2 | 3 | 0.1250 | X.XXX | x.xxx | XX.XXXX |
| | | | Visit 2 | 4 | 0.2500 | x.xxx | x.xxx | XX.XXXX |
| | | | Visit 2 | 5 | 0.5000 | X.XXX | X.XXX | XX.XXXX |
| | | | Visit 2 | 6 | 1.0000 | X.XXX | x.xxx | XX.XXXX |
| | | | Visit 2 | 7 | 2.0000 | X.XXX | x.xxx | XX.XXXX |
| | | | Visit 2 | 8 | 4.0000 | X.XXX | x.xxx | XX.XXXX |
| | | | Visit 2 | 9 | 8.0000 | X.XXX | x.xxx | XX.XXXX |
| | | | Visit 2 | 10 | 16.0000 | X.XXX | x.xxx | XX.XXXX |

#### Protocol / Study No. AI CLR 17 08/ **Albuterol Sulfate Inhalation Aerosol** Visit 2 11 32.0000 X.XXX X.XXX XX.XXXX Visit 2 12 64.0000 X.XXXX.XXX XX.XXXX Visit 2 13 128.0000 X.XXXX.XXX XX.XXXX Visit 2 14 Recovery X.XXXX.XXX XX.XXXX

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

Visit 3 Visit 4 Visit 5

Visit 3-5 will be the same as Visit 2.

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. AI CLR 17 08/

# L16.2.6.3 Listing of Spirometry Test

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Visit | Is the Qualifying FEV <sub>1</sub> >= 80% Predicted Value? / and within 88-112% of Qualifying FEV <sub>1</sub> from the Screening Visit? | Was a 2-Minute Inhalation of a Normal Sterile Saline Control Administered? | Was the Post-saline FEV <sub>1</sub> <= a 10% Drop from the Qualifying FEV <sub>1</sub> and >=70% of Predicted Value? |
|---|---|---|---|---|---|---|
| XX-XXXX | XX-XXXXX | 1 | Visit 2 | Yes | Yes | Yes |
| | | | Visit 3 | Yes | Yes | Yes |
| | | | Visit 4 | Yes | Yes | Yes |
| | | | Visit 5 | Yes | Yes | Yes |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.7.1 Listing of Adverse Events (Safety Population Randomization Period)

| Treatment | Patient<br>Randomi-<br>zation<br>Number | System Organ Class /<br>MedDRA Term /<br>AE Term | Start /End<br>Date | Severity | Relationship<br>to Study<br>Drug | Outcome | Action<br>Taken | Other<br>Action<br>Taken | SAE? |
|---|---|---|---|---|---|---|---|---|---|
| Treatment A | XX-XXXXX | Nervous system disorders /<br>Headache /<br>Headache | yyyy-mm-dd /<br>yyyy-mm-dd | Mild | Possible | Recovered | Dose Not<br>Changed | None | No |
| Treatment B | | | | | | | | | |
| Treatment C | | | | | | | | | |
| Treatment D | | | | | | | | | |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.7.2 Listing of Adverse Events (Safety Population Screening Period)

| Patient<br>Screen<br>Number | System Organ Class /<br>MedDRA Term /<br>AE Term | Start /End<br>Date | Severity | Relationship<br>to Study<br>Drug | Outcome | Action<br>Taken | Other<br>Action<br>Taken | SAE? |
|---|---|---|---|---|---|---|---|---|
| xx-xxxx | Nervous system disorders / | yyyy-mm-dd / | Mild | Possible | Recovered | Dose Not | None | No |
| | Headache / | yyyy-mm-dd | | | | Changed | | |
| | Headache | | | | | | | |

Created on: ddmmmyy hh:mm

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.7.3 Listing of Positive Pregnancy Test Results

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Visit | Results |
|---|---|---|---|---|
| xx-xxxx | XX-XXXXX | 1 | Visit 3 | Positive |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.7.4 Listing of Abnormal Physical Examinations

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Visit | Body<br>System | Result |
|---|---|---|---|---|---|
| xx-xxxx | XX-XXXXX | 1 | Visit 1 | XXXXXXX | Abnormal (xxxxx) |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.8.1 Listing of Vital Signs

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Visit | Time Point | Systolic BP (mmHg) | Diastolic BP (mmHg) | Pulse Rate<br>(beats/min) | Respiration<br>Rate<br>(breaths/min) | Temperature (F) |
|---|---|---|---|---|---|---|---|---|---|
| xx-xxxx | XX-XXXXX | 1 | Visit 1 | Pre-Challenge | 120 | 70 | 84 | 18 | 98.6 |
| | | | | Post-Challenge | 140 | 80 | 74 | 18 | 97.0 |
| | | | Visit 2 | Pre-Challenge | 140 | 80 | 74 | 18 | 97.0 |
| | | | | Post-Challenge | 140 | 80 | 74 | 18 | 97.0 |
| | | | Visit 3 | Pre-Challenge | 140 | 80 | 74 | 18 | 97.0 |
| | | | | Post-Challenge | 140 | 80 | 74 | 18 | 97.0 |
| | | | Visit 4 | Pre-Challenge | 140 | 80 | 74 | 18 | 97.0 |
| | | | | Post-Challenge | 140 | 80 | 74 | 18 | 97.0 |
| | | | Visit 5 | Pre-Challenge | 140 | 80 | 74 | 18 | 97.0 |
| | | | | Post-Challenge | 140 | 80 | 74 | 18 | 97.0 |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

# Protocol / Study No. AI CLR 17 08/

# L16.2.8.2 Listing of 12-Lead ECG

| Patient<br>Screen<br>Number | Patient<br>Randomization<br>Number | Sequence | Visit | ECG<br>Date | ECG<br>Time | ECG<br>Result | Comments |
|---|---|---|---|---|---|---|---|
| xx-xxxx | xx-xxxxx | 1 | Visit 1 | yyyy-mm-dd | hh:mm | Abnormal (Not Clinically Significant) | xxxxxxxxxxxxxxxx |

Sequence: 1=ABCD, 2=DCBA, 3=CADB, 4=BDAC

#### **Albuterol Sulfate Inhalation Aerosol**

Protocol / Study No. AI CLR 17 08/

#### **REFERENCES**

- 1. American Thoracic Society Guidelines for Methacholine and Exercise Challenge Testing. American journal of respiratory and critical care medicine 161, 309-329 (1999).
- 2. Saluja B, D. R., Kim SH, Lee SL. in Respiratory Drug Delivery. 413-416.
- 3. Draft Guidance on Orlistat. Food and Drug Administration's Office of Generic Drugs. Recommended Feb 2010, Revised Aug 2010. Retrieved on Jan 15 2018 from:
  - http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM201268.pdf
- 4. Draft Guidance on Albuterol Sulfate. Food and Drug Administration's Office of Generic Drugs. Recommended Apr 2013, Revised Dec 2016. Retrieved on Jan 15 2018 from: https://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM346985.pdf
- 5. Inman MD, Hamilton AL, Kerstjens HAM, Watson RM, O'Byrne PM. *The utility of methacholine airway responsiveness measurements in evaluating anti-asthma drugs*. J Allergy Clin Immunol. 1998;101(3):342-348
- 6. Mauger EA, Mauger DT, Fish JE, Chinchili VM, Israel E. *Summarizing Methacholine Challenges in Clinical Research*. Control Clin Trials. 2001;22(6 Suppl):244S-251S
- 7. Efron B, Tibshirani RJ. An Introduction to the Bootstrap. (Chapman & Hall: New York, NY, 1993)
- 8. Gibaldi M, Perrier D. Pharmacokinetics, Second Edition, Revised and Expanded. (Marcel Dekker Inc: New York, NY, 1982)
- 9. Bonate PL. Pharmacokinetic-Pharmacodynamic Modeling and Simulation, Second Edition. (Springer Science+Business Media, Inc: New York, NY, 2011)
- 10. StatLib, Department of Statistics, Carnegie Mellon University (http://lib.stat.cmu.edu)

#### NOTE TO FILE

STUDY TITLE: A Randomized, Single-Dose, Double-Blind, Double-Dummy, Four-Period, Four-Sequence, Four-Treatment, Placebo and Active Controlled, Comparative, Multiple-Center, Crossover-Design, Bronchoprovocation Study to Evaluate the Pharmacodynamic Equivalence of Albuterol Sulfate Inhalation Aerosol, eq 90 mcg base (Sun Pharmaceuticals Industries Limited) to PROAIR® HFA (albuterol sulfate) Inhalation Aerosol, eq 90 mcg base (Teva Respiratory, LLC) in Subjects With Stable, Mild Asthma

**PROTOCOL NO.:** CLR 17 08 (Revision 6.0)

This Note to File explains the changing of numbering as per ICH guidance E3 for Tables, Listings and Figures that are included in the final SAP dated December 21, 2018.

- T14.1.1 Summary of Patient Disposition
- T14.1.2 Summary of Protocol Deviations
- T14.1.3 Summary of Patient's Treatments Included in the Pharmacodynamic Analysis
- T14.1.4 Summary of Demographic Data and Baseline Characteristics
- T14.1.5 Summary of Demographic Data and Baseline Characteristics
- T14.1.6 Summary of Demographic Data and Baseline Characteristics
- T14.2.1.1 Summary of Concentration (mg/mL) of Methacholine Required to Reduce FEV<sub>1</sub> by 20% (PC<sub>20</sub>) (Safety Population)
- T14.2.1.2 Summary of Concentration (mg/mL) of Methacholine Required to Reduce FEV<sub>1</sub> by 20% (PC<sub>20</sub>) (Pharmacodynamic Population)
- T14.2.1.3 Summary of Concentration (mg/mL) of Methacholine Required to Reduce FEV<sub>1</sub> by 20% (PC<sub>20</sub>) (Per-Protocol Population)
- T14.2.2.1 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 second ( $FEV_1$ ) (Safety Population)
- T14.2.2.2 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 second ( $FEV_1$ ) (Pharmacodynamic Population)
- T14.2.2.3 Summary of Pre-challenge Forced Expiratory Volume (flow rate) in 1 second ( $FEV_1$ ) (Per-Protocol Population)
- T14.3.1.1 Overall Summary of Adverse Events
- T14.3.1.2 Summary of Frequency of All Adverse Events by System Organ Class
- T14.3.1.3 Summary of Frequency of Serious Adverse Events by System Organ Class
- T14.3.1.4 Summary of Frequency of All Adverse Events by Relationship to Study Drug
- T14.3.1.5 Summary of Frequency of Serious Adverse Events by Relationship to Study Drug
- T14.3.1.6 Summary of Frequency of All Adverse Events by Severity

- T14.3.1.7 Summary of Frequency of Serious Adverse Events by Severity
- T14.3.2 Summary of Vital Signs
- L16.2.1.1 Listing of Discontinued Subjects
- L16.2.2.1 Listing of Protocol Deviations
- L16.2.3.1.1 Listing of Subjects Excluded from the Per-Protocol Population
- L16.2.3.1.2 Listing of Subjects Excluded from the Per-Protocol Population for analysis
- L16.2.3.2 Listing of Subjects Excluded from the Pharmacodynamic Population
- L16.2.4.1 Listing of Demographic Data
- L16.2.4.2 Listing of Medical History
- L16.2.5.1 Listing of Concomitant Medication
- L16.2.5.2 Listing of Dosing
- L16.2.6.1 Listing of Methacholine Challenge and Pulse Oximetry
- L16.2.6.2 Listing of Methacholine Challenge Stages
- L16.2.6.3 Listing of Spirometry Test
- L16.2.7.1 Listing of Adverse Events (Safety Population Randomization Period)
- L16.2.7.2 Listing of Adverse Events (Safety Population Screening Period)
- L16.2.8.1 Listing of Positive Pregnancy Test Results
- L16.2.8.2 Listing of Abnormal Physical Examinations
- L16.2.8.3 Listing of Vital Signs
- L16.2.8.4 Listing of 12-Lead ECG

